CLINICAL TRIAL: NCT03860311
Title: BULLET: Bladder Ultrasound Limits Length (of Time), Expedites Treatment
Acronym: BULLET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Stephen Ruffenach, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB-300002071
Record Dates: First submitted 2019-02-28; First posted 2019-03-01 (Actual); Results first posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Point-of-Care Bladder Ultrasound; Urethral Catheter
Keywords: Ovarian Torsion; Point-of-Care; Pelvic pain; Bedside Ultrasound
MeSH Terms: conditions — Ovarian Torsion; Pelvic Pain | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Bladder Ultrasound (Experimental): The bladder ultrasound group will undergo point-of-care ultrasound upon enrollment, and bladder ultrasound will be repeated every 30 minutes, unless the patient's bladder is full at time of initial scan.
  Interventions: Device: Bladder Ultrasound
- Standard of Care (Active Comparator): Bladder (Urethral) Catheter group. The standard of care group will undergo placement of a urethral bladder catheter to allow retrograde filling of the bladder.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: Bladder Ultrasound — Bladder fullness will be assessed upon enrollment and if not full, the patient will receive hydration, determined by treating physician, and the bladder ultrasound will be repeated every 30 minutes until the patient states that the bladder is "full," or until bladder is deemed full based on a previously validated bladder fullness qualitative scale, at which point patients in this group will proceed to undergo pelvic ultrasound.
  Arms: Bladder Ultrasound
Other: Standard of Care — Per institution protocol, patients in the standard of care group will have urethral (bladder) catheter placed immediately after the order for pelvic ultrasound and will undergo retrograde bladder filling as determined by the radiologist/ultrasonographer to the point necessary to fully visualize pelvic structures.
  Arms: Standard of Care

SUMMARY:
In this study patients presenting to the pediatric ER with abdominal or pelvic complaints will be randomized to urethral bladder catheter or bladder ultrasound to compare time to completion of successful pelvic ultrasound, as determined by full visualization of uterus and ovaries.

DETAILED DESCRIPTION:
In this study, we will enroll female pediatric emergency department (ED) patients presenting with a diagnosis of abdominal pain who may have a transabdominal pelvic ultrasound ordered by their treating physician (or nurse practitioner). In order to maximize the visualization of organs deep within the pelvis such as the ovaries and uterus, the patient's bladder must be full. The current practice at our institution, as well as numerous others, is to have a bladder catheter placed immediately when a transabdominal pelvic ultrasound is ordered, and then to fill the bladder in a retrograde manner in order to provide enhanced visualization of the pelvic structures. The process of inserting a bladder catheter into a pediatric patient is an invasive procedure which can be traumatic and painful to the patient. Additionally, if the patient's bladder is already full, this procedure may be unnecessary.

In this study, a point-of-care bladder ultrasound will be performed, upon enrollment of a patient by a study bedside sonographer (our pediatric emergency department nurse practitioners), to assess degree of bladder fullness. This measurement will then be repeated serially while the patient is receiving hydration and the ultrasound will be performed when the bladder is full. We hypothesize that this work flow will result in an equivalent time to transabdominal pelvic ultrasound completion and will reduce the number of potentially traumatic and painful, invasive urethral bladder catheterizations.

ELIGIBILITY:
Inclusion Criteria:

* Age 8yr-18yrs
* Female
* Likely to have order placed for transabdominal pelvic ultrasound/ovarian ultrasound
* No history of pelvic or bladder reconstructive surgery

Exclusion Criteria:

* Pregnancy (known)
* Critically ill patients
* Patients with known renal or genitourinary structural abnormalities or prior pelvic/genitourinary surgery
* Chronic renal disease
* Patients presenting outside the defined treatment windows

Ages: 8 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Participants will be females visiting the emergency department for abdominal, vaginal, or possible genitourinary-related complaints, which may include abdominal pain, vaginal discharge, pelvic bleeding, flank pain, or vomiting, and for which treating physicians have a concern for pelvic pathology, such as ovarian torsion, ovarian cysts, or other ovarian or uterine pathology.
Enrollment: 45 (Actual)
Dates: Start 2019-07-20 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen R Richard, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bladder Ultrasound | Standard of Care
Started | 22 | 23
Completed | 22 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bladder Ultrasound | Standard of Care | Total
Number analyzed (Participants) | 22 | 23 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.33 (1.98) | 14.7 (2.183) | 15.00 (2.091)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 45
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 5 | 12
  White | 14 | 17 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 22 | 23 | 45

OUTCOME MEASURES:

1. Primary Outcome: Time to Successful Completion of Pelvic Ultrasound
Description: Time zero (order placed) to time completed (time pelvic ultrasound images are completed)
Time Frame: Baseline to 180 minutes
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Bladder Ultrasound | Standard of Care
Number analyzed (Participants) | 22 | 23
minutes | 103.95 [82.64 to 125.27] | 92.82 [80.29 to 105.35]

2. Secondary Outcome: Pain of Bladder Ultrasound vs. Pain of Bladder Catheter as Measured by Verbal Numerical Rating Scale (VNRS)
Description: All participating patients, in either arm, will be given a single-question on pain related to their receipt of bladder ultrasound(s) or bladder catheter. The VNRS uses a 0-10 scale accompanied by faces that pictorially represent the level of pain, 0 being no pain, and 10 being the worst pain. Measurements will start at time when bladder ultrasound(s) are performed OR time when bladder catheter is inserted) to time of completion (time pelvic ultrasound is completed).
Time Frame: When bladder ultrasound performed OR when urinary catheter placed to time of completion of pelvic ultrasound, up to 180 minutes
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Bladder Ultrasound | Standard of Care
Number analyzed (Participants) | 22 | 23
units on a scale | 3.60 [2.14 to 5.06] | 6.23 [5.40 to 7.06]

ADVERSE EVENTS:
Time Frame: The time the patient remained in the emergency department (172mins-921mins)
Arm/Group | Bladder Ultrasound | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/23
Other Adverse Events (participants affected / at risk) | 0/22 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-02-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT03860311/Prot_000.pdf